CLINICAL TRIAL: NCT05566730
Title: Mobile App to Address CUD Among Black Adults
Brief Title: Culturally Tailored Cannabis Use Disorder App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Louisiana State University Health Sciences Center in New Orleans (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Lorra Garey, Principal Investigator, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003690; U54MD015946 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-10-04 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cannabis Use
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-MICART App (Experimental): Participants in this arm will receive daily EMAs for 6 weeks.
  Interventions: Behavioral: CT-MICART App; Behavioral: Control

INTERVENTIONS:
Behavioral: CT-MICART App — App designed with the goal of treating CUD in African American adults
Behavioral: Control — App designed with the goal of treating CUD in African American adults, with participants just tracking their use of cannabis and not receiving treatment videos
  Other Names: Sham

SUMMARY:
The present study aims to address disparities in cannabis use outcomes among African American/Black (hereby referred to as Black) adults with cannabis use disorder (CUD). The specific aims of this study are: (1) to develop a culturally adapted, mobile app for Black cannabis users (CT-MICART) using knowledge from the current research team, published literature, expert opinion, and feedback from the Community Research Advisory Board (CRAB), (2) to pilot test CT-MICART and (3) focus on analysis of data collected as part of Aim 2.

DETAILED DESCRIPTION:
The present study aims to address disparities in cannabis use outcomes among African American/Black (hereby referred to as Black) adults with cannabis use disorder (CUD). African American/Black adults are more likely to endorse cannabis use patterns that are more severe (weekly and blunt use) and meet diagnostic criteria for cannabis use disorder (CUD) than White adults (16.8% vs 10.0%). This finding is alarming as cannabis use disorder is associated with more severe psychosocial risk profiles, including poly-substance use, psychiatric problems, and legal trouble relative to non-CUD use and non-use. Additionally, although Black cannabis users are more likely to report being ready to quit and a recent quit attempt relative to White cannabis users, this population is less likely to seek in-person treatment relative to White cannabis users because of individual (e.g., beliefs about use), community (e.g., neighborhood attitudes about use), and institutional (e.g., healthcare access) factors as well as due to institutionalized racism and discrimination (e.g., more likely to not be listened to by practitioners). Targeted, accessible, and culturally adapted therapeutic programming is needed to reduce risk and improve disparities for poor cannabis-related outcomes among Black adults with cannabis use disorder. These findings are significant because they contribute to heath, social, and psychological health disparities within the Black community. Psycho-sociocultural models of substance use posit that Black individuals may use cannabis and continue using despite cannabis-related problems including cannabis use disorder, to manage psychological distress associated with stressors associated with minority status, such as racial discrimination. Therefore, the present study seeks to develop a culturally adapted, mobile app tailored specifically for Black cannabis users (CT-MICART). Using the expert opinion and feedback from the community Research Advisory Board (CRAB), the investigative team will pilot test CT-MICART and focus on analysis of data collected to help achieve a better culturally tailored app.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* identify as Black/African American
* CUD per CUPIT-R
* willing and able to complete study appointments
* motivated to reduce cannabis (≥5 on a 10-point scale)
* score ≥ 4 on the REALM-SF indicating ≥ 6th grade English literacy level (needed to use app)
* report cannabis use to manage anxiety/stress in the past month

Exclusion Criteria:

* legal mandate or substance misuse treatment
* report of current or intended participation in a concurrent substance use treatment, including pharmacotherapy or psychotherapy for CUD not provided by researchers
* ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety or depression
* not being fluent in English
* pregnant of planning to become pregnant within the next six months (assessed via self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Safety Aid Scale | Baseline appointment and 6-week follow up appointment
  The Safety Aid Scale will be used to assess change of false safety behavior use over time, being scored on a 5 point scale where higher scores indicate greater use of false safety behaviors.
Qualitative Interview | 6-week follow up appointment
  The qualitative interview done by the participants will ask them about their experience with the app, what aspects helped, what aspects didn't help, and will allow researchers to adapt and refine the CT-MICART app.
Engagement with the CT-MICART app | Week 1-6
  Behavioral indicators of engagement with the app (>75% of all videos watched and >75% of scheduled skills practiced).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Nizio P, Clausen B, Businelle MS, Ponton N, Jones AA, Redmond BY, Buckner JD, Obasi EM, Zvolensky MJ, Garey L. Mobile Intervention to Address Cannabis Use Disorder Among Black Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 19;13:e52776. doi: 10.2196/52776. PMID 38373037